CLINICAL TRIAL: NCT06549998
Title: Effects of High-Fidelity Patient Simulation on Clinical Reasoning Skills and Interprofessional Competencies in Physical Therapy and Nursing Students
Brief Title: High-Fidelity Patient Simulation on Clinical Reasoning Skills and Interprofessional Competencies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Youngstown State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2024-260
Record Dates: First submitted 2024-08-05; First posted 2024-08-12 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: nursing; physical therapy; education; interprofessional; simulation; clinical reasoning

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): This group will not receive any simulation intervention
- Experimental Group (Experimental): This group will receive 2 simulations
  Interventions: Other: Interprofessional Simulation Experience

INTERVENTIONS:
Other: Interprofessional Simulation Experience — Phase 1 (Pre-Brief): Nursing and physical therapy students will have 10 minutes to gather as a group and prepare for the simulation experience.
  The students will work together to review the simulated patient's medical chart, which includes a hand off report, physician orders, patient demographic data, disci-pline-specific progress notes, a physical therapy evaluation, and information from lab results posted on a tri-fold board.
  Phase 2 (Simulation): After reviewing the chart and establishing a plan as a group for getting the simulated patient out of bed, the interprofessional team of nursing and physical therapy students will enter the simulated hospital room. The goal for the approximately 20-minute encounter is for the interprofessional group to help the simulated patient to get out of bed while closely monitoring the physiological responses to activity.
  Phase 3: The simulation will conclude with a 30-minute faculty guided and structured debriefing session.
  Arms: Experimental Group

SUMMARY:
The proposed study is looking to examine the effects of High-Fidelity Patient Simulation (HFPS) on clinical reasoning skills and interprofessional competencies in Physical Therapy and Nursing students.

The proposed study will have two objectives:

1. Assess the use of HFPS and whether it has an effect of improving physical therapy and nursing student performance related to clinical reasoning skills during simulated clinical situations.
2. Assess the use of HFPS and whether it has an effect of improving physical therapy and nursing student self-reported changes in team work and communication based on the IPEC core competencies

Researchers will compare students who do not receive a simulation (Group C) to those who receive two simulations (Group E).

Participants will:

1. Be assigned to one of 2 groups (Group C, Group E)
2. Based on group assignment receive no simulation or 2 simulations
3. Each group will be assessed at the end for their inter-professional attitudes and clinical reasoning skills

DETAILED DESCRIPTION:
Background Information Patient-centered care is important in helping individuals who live with multiple health conditions, requiring collaboration among healthcare professionals of different disciplines. Interprofessional collaborative practice has been defined by the World Health Organization as "multiple health workers from different professional backgrounds working together with patients, families, caregivers, and communities to deliver the highest quality of care". It is difficult for any one healthcare professional to address the number and variety of healthcare problems, making collaboration an important part of healthcare. An ability to effectively collaborate among health care disciplines in the areas of communication, role identification, team working skills, and conflict resolution are critical components of practice for health care professionals. This has led to educational institutions placing a greater emphasis on the development and integration of interprofessional education (IPE) into health professions curricula. The emphasis of IPE is to prepare health professions students to work together with the aim of building a safe, patient-centered health care environment5.

Experiential learning provides learners an opportunity to practice skills and techniques learned in the classroom in a real-world or practical setting. The benefits of experiential learning have long been held in high regard and include enhancing understanding of content and improvement in interpersonal skills. Implementation of experiential learning varies significantly across PT curricula. Some experiential learning methods are time and labor intensive, while others are less so. Cost, feasibility, time constraints, and course outcomes play a role in determining which methods work best for a particular course or program. Simulation has been used for decades to assist with skill acquisition and assessment. High-fidelity human patient simulation (HFPS) with a focus on clinical situations/scenarios is highly conducive to IPE. The term "simulation" refers to an experiential educational technique which "creates a situation or environment to allow persons to experience a representation of a real event for the purpose of practice, learning, evaluation, testing, or to gain understanding of systems or human actions.". In health care simulation, high-fidelity refers to "simulation experiences that are extremely realistic and provide a high level of interactivity and realism for the learner".

The use of simulation as a teaching pedagogy can be especially valuable in replicating the acute care setting.

Statement of the Problem The Interprofessional Education Collaborative (IPEC) set forth a series of core competencies for interprofessional collaborative practice. The IPEC describes these core competencies as: " to the safe, high-quality, accessible, patient-centered care and enhanced population health outcomes desired by all". These core competencies were developed in order to prepare students to engage in lifelong learning and collaboration to improve community health outcomes. These competencies include: Values and Ethics (work with team members to maintain a climate of shared values, ethical conduct, and mutual respect), Roles and Responsibilities (Use the knowledge of one's own role and team members' expertise to address health outcomes), Communication (Communicate in a responsive, responsible, respectful, and compassionate manner with team members.), Teams and Teamwork (Apply values and principles of team science to adapt one's own role in a variety of team settings).

The use of HFPS has been utilized in education settings involving physical therapy students. A recent review that examined the effect of HFPS learning in Acute Cardiorespiratory Physical Therapy noted that there is currently a lack of quality studies that have examined this area of study. Part of the quality involved the choice of research design and the lack of validated outcome measures to assess variables of interest. The review was unable to determine whether HFPS can improve physical therapists' clinical performance and/or preparedness. In addition, many studies examine pre-post simulation when capturing outcome data, demonstrating a further need for longer longitudinal studies to further assess student performance. There is also reported variability in how HFPS is used, the optimal delivery, timing, volume, and content.

The proposed study will have two objectives:

1. Assess the use of HFPS and whether it has an effect of improving physical therapy and nursing student performance related to clinical reasoning skills during simulated clinical situations.
2. Assess the use of HFPS and whether it has an effect of improving physical therapy and nursing student self-reported changes in team work and communication based on the IPEC core competencies.

ELIGIBILITY:
Inclusion Criteria:

- Must be a student currently enrolled in either the physical therapy or nursing program

Exclusion Criteria:

- Not currently enrolled as a student in the physical therapy or nursing program

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-05-17 (Actual); Study Completion 2025-05-17 (Actual)

PRIMARY OUTCOMES:
Interprofessional Attitudes Scale (IPAS) | baseline and through study completion (an average of 8 months)
  The tool measures 5 subscales that include: Teamwork roles and responsibilities, Patient centeredness, Interprofessional biases, Diversity and ethics, Community centeredness. The IPAS is based off of the 4 competencies for interprofessional education.
  The tool is a 27 item 5-point agreement scale ranging from strongly disagree to strongly agree. Internal consistency reliability for the sub-scales were good (i.e., Cronbach alpha = 0.62 to 0.92). Exploratory factor analysis revealed that items loaded sufficiently (i.e., loading greater than 0.30) on only one of five factors (i.e., did not cross-load). Confirmatory factor analysis supported the sub-scale structure, Goodness of Fit Index (GFI) = 0.86 and Root Mean Squared Error of Approximation (RMSEA) = 0.90.
Lasater Clinical Judgment Rubric (LCJR) | baseline and through study completion (an average of 8 months)
  The rubric's 11 dimensions of student performance are grouped into 4 subscales (Noticing, Interpreting, Responding, and Reflecting), with clear performance descriptions for dimension scores between 1 (beginning) and 4 (exemplary), and LCJR totals between 11 and 44 points. The LCJR is considered a valid and reliable instrument with the Cronbach α for total scores between 0.80 and 0.97 and subscale results of 0.89 to 0.93. Although it has been mainly used in simulation, use of the LCJR in clinically focused studies has been successful with Manetti reporting reliability of 0.89.
Performance Assessment Communication and Teamwork Tool Set (PACT) | baseline and through study completion (an average of 8 months)
  The PACT tools are designed to provide assessment feedback for learners, and evaluation information for program faculty. For this study, only the expert observation rating tool will be used. The overall inter-rater reliability of the novice, expert, and video observational tools was good (Intraclass Correlation Coefficient (ICC) = 0.85, 0.76, and 0.90, respectively). The inter-rater reliability for four of the five domains in the expert observational tool were acceptable (ICC = 0.44-0.66); the exception was the team structure domain (ICC = 0.21). The inter-rater reliability for all five domains in the video observational tool were acceptable (ICC = 0.54-0.84).

CONTACTS AND LOCATIONS:
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States

REFERENCES:
- [Background] Nandan M, Scott PA. Interprofessional practice and education: holistic approaches to complex health care challenges. J Allied Health. 2014 Aug;43(3):150-6. PMID 25194061
- [Background] Nichols A, Wiley S, Morrell BL, Jochum JE, Moore ES, Carmack JN, Hetzler KE, Toon J, Hess JL, Meer M, Moore SM. Interprofessional Healthcare Students' Perceptions of a Simulation-Based Learning Experience. J Allied Health. 2019 Fall;48(3):159-166. PMID 31487353
- [Background] Bethea DP, Smith N, Allison LK, Bell CS, Collins ME, Migliarese SJ, Darby R. Live Standardized Patient Scenario Improves Attitudes Toward and Readiness for Interprofessional Education in Occupational Therapy and Physical Therapy Students. J Allied Health. 2019 Summer;48(2):81-87. PMID 31167008
- [Background] Smith SN, Crocker AF. Experiential learning in physical therapy education. Adv Med Educ Pract. 2017 Jun 28;8:427-433. doi: 10.2147/AMEP.S140373. eCollection 2017. PMID 28721117
- [Background] Rossler KL, Kimble LP. Capturing readiness to learn and collaboration as explored with an interprofessional simulation scenario: A mixed-methods research study. Nurse Educ Today. 2016 Jan;36:348-53. doi: 10.1016/j.nedt.2015.08.018. Epub 2015 Sep 1. PMID 26363963
- [Background] Blaseg NA. Simulation-Based Interprofessional ICU Bedside Rounding Course. S D Med. 2022 Oct;75(10):449-450. PMID 36889260
- [Background] Coppola AC, Coppard BM, Qi Y. Impact of Participation in an Interprofessional Acute Care High-Fidelity Simulation for Occupational and Physical Therapy Graduate Students. J Allied Health. 2019 Winter;48(4):248-256. PMID 31800654
- [Background] Karnish K, Shustack L, Brogan L, Capitano G, Cunfer A. Interprofessional Socialization Through Acute-Care Simulation. Radiol Technol. 2019 Jul;90(6):552-562. PMID 31270256
- [Background] Shoemaker MJ, Riemersma L, Perkins R. Use of high fidelity human simulation to teach physical therapist decision-making skills for the intensive care setting. Cardiopulm Phys Ther J. 2009 Mar;20(1):13-8. PMID 20467529
- [Background] Silberman NJ, Panzarella KJ, Melzer BA. Using human simulation to prepare physical therapy students for acute care clinical practice. J Allied Health. 2013 Spring;42(1):25-32. PMID 23471282
- [Background] Thomas EM, Rybski MF, Apke TL, Kegelmeyer DA, Kloos AD. An acute interprofessional simulation experience for occupational and physical therapy students: Key findings from a survey study. J Interprof Care. 2017 May;31(3):317-324. doi: 10.1080/13561820.2017.1280006. Epub 2017 Feb 28. PMID 28276844
- [Background] Wellmon R, Lefebvre KM, Ferry D. Effects of High-Fidelity Simulation on Physical Therapy and Nursing Students' Attitudes Toward Interprofessional Learning and Collaboration. J Nurs Educ. 2017 Aug 1;56(8):456-465. doi: 10.3928/01484834-20170712-03. PMID 28787067